CLINICAL TRIAL: NCT00864084
Title: Does a Pulmonary Rehabilitation Program Improve Balance in Individuals With Respiratory Disease?
Brief Title: Does Pulmonary Rehabilitation Improve Balance in People With Respiratory Disease?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Ms. Elizabeth Harvey, Ms, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2009:007
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): People with respiratory disease
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pulmonary rehabilitation involves the prescription of customized exercise programs and education on disease management.

SUMMARY:
The purpose of this study is to determine whether participation in pulmonary rehabilitation improves balance in people with respiratory disease.

DETAILED DESCRIPTION:
Falls and chronic respiratory are two major health concerns affecting morbidity and mortality in older adults. Several factors that predispose falls, such as reduced balance, have been documented in people with respiratory disease. Pulmonary rehabilitation programs, which involve customized exercise prescription, are recommended to improve quality of life and disease management in people with chronic obstructive pulmonary disease (COPD). There are many documented benefits to participation in such programs; however, the impact on balance and other falls risk factors has not previously been investigated. Therefore, the aim of this study is to investigate the effect of a pulmonary rehabilitation program on balance and falls risk factors in individuals with respiratory disease. This study will enhance the current management of respiratory disease by improving our understanding of the effects of pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lung disease
* Committed to regular attendance at pulmonary rehabilitation program
* A forced expiratory volume in 1 second (FEV1) < 80% of predicted
* No change in medications for the past 2 months

Exclusion Criteria:

* Unstable cardiac disease
* Neurological conditions
* Musculoskeletal conditions that prevent participation in exercise sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle D Smith, PhD, Principal Investigator — The University of Queensland
Locations (1):
- The University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Smith MD, Harvey EH, van den Hoorn W, Shay BL, Pereira GM, Hodges PW. Out-Patient Pulmonary Rehabilitation Improves Medial-Lateral Balance in Subjects With Chronic Respiratory Disease: Proof-of-Concept Study. Respir Care. 2016 Apr;61(4):510-20. doi: 10.4187/respcare.04109. Epub 2016 Jan 26. PMID 26814219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven individuals with stable chronic respiratory disease who were attendees of an institutional outpatient pulmonary rehabilitation program participated in this study. Recruitment occurred in April 2009 and at the pulmonary rehabilitation program.
Pre-assignment Details: People enrolled in the pulmonary rehabilitation programs who had a clinical diagnosis of respiratory disease were included in the study. Exclusion criteria were: unstable cardiac disease, neurological conditions, or musculoskeletal conditions that prevented participation in pulmonary rehabilitation or testing sessions.
Groups:
- Pulmonary Rehabilitation: An 8-week out-patient pulmonary rehabilitation program.
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pulmonary Rehabilitation
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  Canada | 14

OUTCOME MEASURES:

1. Primary Outcome: Standing Balance - Sway Path
Description: Standing balance was measured using a force plate (AMTI, Watertown, MA, USA) from which centre of pressure (COP) trajectories were derived at a sampling frequency of 100Hz. Participants stood on the force plate during the following two conditions: normal stance (feet hip-width apart) with eyes open and eyes closed.
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Pre-pulmonary Rehabilitation - Eyes Open; Post-pulmonary Rehabilitation - Eyes Open: Participant data prior to participation in an 8-week outpatient pulmonary rehabilitation program. Standing balance testing by standing on the force plate with eyes open.
- Pre-pulmonary Rehabilitation - Eyes Closed; Post-pulmonary Rehabilitation - Eyes Closed: Participant data prior to participation in an 8-week outpatient pulmonary rehabilitation program. Standing balance testing by standing on the force plate with eyes closed.
Arm/Group | Pre-pulmonary Rehabilitation - Eyes Open | Pre-pulmonary Rehabilitation - Eyes Closed | Post-pulmonary Rehabilitation - Eyes Open | Post-pulmonary Rehabilitation - Eyes Closed
Number analyzed (Participants) | 11 | 11 | 11 | 11
cm/s
  Anteroposterior sway path | 1.57 (0.91) | 3.40 (3.10) | 1.65 (0.61) | 2.59 (1.68)
  Mediolateral sway path (cm/s) | 0.60 (0.35) | 1.22 (0.90) | 0.67 (0.36) | 0.79 (0.43)

2. Primary Outcome: Dynamic Balance
Description: Dynamic balance was measured using the timed up and go (TUG) and Four Square Step Test (FSST). For the TUG, the time taken for the subject to stand from a chair, walk 3 m, turn around and return to the chair was recorded {Podsiadlo, 1991 #31}. Subjects were asked to do this as quickly and safely as possible. High test-retest reliability of the TUG has been reported in older community-dwelling individuals {Steffen, 2002 #34}. In the FSST, subjects were asked to step to four corners of a square in a clockwise and then counter-clockwise direction as quickly as possible {Dite, 2002 #1181}. The time taken to complete this circuit was recorded. This test has been shown to have high inter-rater and test-retest reliability {Dite, 2002 #1181}.
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Pre-pulmonary Rehabilitation: Participant data prior to participation in an 8-week outpatient pulmonary rehabilitation program.
- Post-pulmonary Rehabilitation: Participant data after participation in an 8-week outpatient pulmonary rehabilitation program.
Arm/Group | Pre-pulmonary Rehabilitation | Post-pulmonary Rehabilitation
Number analyzed (Participants) | 11 | 11
seconds
  Timed Up and Go | 10.7 (4.45) | 9.26 (3.36)
  Four Square Step Test | 11.1 (5.03) | 9.23 (2.72)

3. Secondary Outcome: Balance Confidence
Description: Activity-Specific Balance Confidence (ABC) scale measures balance confidence during sixteen activities of progressive difficulty, such as going up and down stairs, reaching for objects and walking in crowded areas {Powell, 1995 #5}. It asks subjects to rate their level of confidence in performing an activity without losing balance on an 11-point scale ranging from 0% (no confidence) to 100% (completely confident). The score is calculated as the average score for each item. This questionnaire has been shown to be sensitive to detect changes in function following rehabilitation {Myers, 1998 #6} and has proven internal consistency and test-retest reliability {Powell, 1995 #5}.
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-pulmonary Rehabilitation | Post-pulmonary Rehabilitation
Number analyzed (Participants) | 11 | 11
units on a scale | 75.3 (20.3) | 72.0 (21.4)

4. Secondary Outcome: Fear of Falling
Description: The Falls Efficacy Scale International (FESI) assesses fear of falling during a range of physical and social activities {Yardley, 2005 #1}. It asks about an individual's concern about the possibility of following during participation in sixteen common activities, such as cleaning the house, ascending and descending stairs and walking in various environmental conditions. Answers range from 1, "not at all" concerned, to 4, "very" concerned, on a 4-point scale, and score is calculated as the average response. This questionnaire has been shown to have excellent internal and test-retest reliability {Yardley, 2005 #1}.
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pre-pulmonary Rehabilitation | Post-pulmonary Rehabilitation
Number analyzed (Participants) | 11 | 11
scores on a scale | 1.78 (0.63) | 1.83 (0.59)

5. Secondary Outcome: Confidence in Disease Management
Description: The COPD Self-Efficacy Scale evaluates level of confidence in ability to manage or avoid breathing difficulty during a range of situations such as feeling frustrated and lifting heavy objects {Wigal, 1991 #3}. Possible answers range from "very confident" (5 points) to "not at all confident" (1 point) and the average score per question is calculated. This scale has been shown to have excellent internal consistency and good test-retest reliability.
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pre-pulmonary Rehabilitation | Post-pulmonary Rehabilitation
Number analyzed (Participants) | 11 | 11
scores on a scale | 3.27 (0.68) | 3.56 (0.71)

6. Primary Outcome: Standing Balance - Critical Point in Time
Description: as for outcome 1
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Pre-pulmonary Rehabilitation - Eyes Open | Pre-pulmonary Rehabilitation - Eyes Closed | Post-pulmonary Rehabilitation - Eyes Open | Post-pulmonary Rehabilitation - Eyes Closed
Number analyzed (Participants) | 11 | 11 | 11 | 11
s
  Anteroposterior critical point in time (s) | 1.17 (0.48) | 0.87 (0.57) | 1.18 (0.71) | 0.81 (0.42)
  Mediolateral critical point in time | 1.26 (0.51) | 1.22 (0.76) | 1.08 (0.21) | 0.95 (0.45)

7. Primary Outcome: Standing Balance - Critical Point in Distance
Description: as for outcome 1
Time Frame: Baseline (pre-pulmonary rehabilitation) and follow-up (post-pulmonary rehabilitation) at 8 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pre-pulmonary Rehabilitation - Eyes Open | Pre-pulmonary Rehabilitation - Eyes Closed | Post-pulmonary Rehabilitation - Eyes Open | Post-pulmonary Rehabilitation - Eyes Closed
Number analyzed (Participants) | 11 | 11 | 11 | 11
cm
  Anteroposterior critical point in distance (cm) | 0.54 (0.34) | 1.36 (1.25) | 0.71 (0.65) | 1.05 (0.84)
  Mediolateral critical point in distance | 0.19 (0.28) | 0.55 (0.67) | 0.21 (0.21) | 0.17 (0.18)

ADVERSE EVENTS:
Groups:
- Study Participation: Participant data collection at baseline (pre-pulmonary rehabilitation), participation in an 8-week outpatient pulmonary rehabilitation program and data collection at follow-up (post-pulmonary rehabilitation).
Arm/Group | Study Participation
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
This sample size in this study was small. Study participants received an individualised exercise program which means that exercises given and number of pulmonary rehabilitation sessions attended were not standardized between study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No